CLINICAL TRIAL: NCT06833554
Title: The Role of Breast Milk Neutrophils From Mothers With Metabolic Diseases and Impact on Infant Development and Response to Pulmonary Infections
Brief Title: The Role of Breast Milk Neutrophils From Mothers With Metabolic Diseases After Nutritional Intervention. Impact on Infant Development and Response to Pulmonary Infections
Acronym: PI2222/01813
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI22/01813
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Gestational Diabetes Mellitus (GDM)
MeSH Terms: conditions — Diabetes, Gestational | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 (Active Comparator)
  Interventions: Dietary Supplement: Omega-3 Fatty Acids (EPA plus DHA)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids (EPA plus DHA) — Dietary supplementation with Omega-3 Fatty Acids to study the effect on the immune system of breast milk
  Arms: Omega-3
Dietary Supplement: Placebo — Inert dietary supplement, without activity in the activation of the immune system of breast milk
  Arms: Placebo

SUMMARY:
This project aims at identifying variations in breast milk neutrophils among lactating mothers with gestational diabetes or obesity (objective 1), and to describe how a dietary intervention with Omega-3 fatty acids affects these changes (objective 2). The occurrence of respiratory infections on the progeny will be analysed, as well as its development and the impact on gut microbiota and epigenetic changes (objective 3). The involvement of breast milk on the neonate's microbiota (sub-objective 1) and epigenetic variations (sub-objective 2) will be depicted. In addition, the direct engagement of milk neutrophils in the ability of the progeny to react against lung infections will be studied (sub-objective 3).

To attain these mother milk and blood samples will be obtained from three groups of lactating mothers: control, obesity or gestational diabetes, upon a dietary intervention with Omega-3 fatty acids. Neutrophil populations of maternal blood and milk samples will be studied by flow cytometry and in vitro assays. The microbiome and miRNA content of infant's saliva and tool samples will be characterized by 16s rRNA gene sequencing and PCR. The occurrence of respiratory infections and the development the infants participating in the study will be tracked during the first 2 years of life by telephone surveys.

To study the impact of the presented maternal variables on the progeny upon a respiratory inflammation on a systemic level, mouse models will be employed. The offspring of lactating dams with gestational diabetes or obesity will be subjected to an artificial acute lung infection. The progression of the lung disease will be studied by histology and the neutrophil profile in the organs of the litter by flow cytometry. The response to acute lung injury after fecal transplantation with infant's microbiota intro germ-free mice as well as of wild type pups breastfeed by neutropenic dams will complement the animal studies.

ELIGIBILITY:
Inclusion Criteria:

* full term pregnancy (>37 weeks)
* mother age 18-50 years
* intention to practice exclusive breastfeeding for at least 3 months

Exclusion Criteria:

* preterm pregnancy (<37 weeks)
* multiple delivery
* delivery complications that compromise the well-being of the newborn
* congenital abnormalities of the baby
* pathologies of the mother such as hypertension, HELLP syndrome, thyroids alterations or nephropathies - drugs or alcohol abuse record
* occurrence of mastitis during the study
* mothers practicing tandem nursing

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female participants are eligible as the study is focused on lactation
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of milk neutrophils from three groups of lactating mothers: control or gestational diabetes. | From enrollment to end of treatment at 3 months
Characterization of microbiota and miRNA content of breast milk | From enrollment to end of treatment at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- IBIMA-Plataforma Bionand, Málaga, Malaga, Spain